CLINICAL TRIAL: NCT01561066
Title: Adjuvant Use of Autologous Platelet-rich Fibrin Glue in the Treatment of Fistulas and Anastomotic Leakages of the Digestive Tract
Brief Title: Autologous Fibrin Glues for Fistulas Closure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Clinical professor, Principal investigator, Jinling Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRA2011232-1
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Enterocutaneous Fistulas; Intra-abdominal Infection
Keywords: Fibrin glue; Platelet; Autologous derivation; Prospective randomized trial; Fistulas
MeSH Terms: conditions — Intestinal Fistula; Intraabdominal Infections; Fistula | interventions — Octreotide; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conservative therapy (Sham Comparator): Conservative therapy includes orrection of electrolytic disturbances, suppression of gastric/intestinal secretion with octreotide, nutritional support.
  Interventions: Drug: Octreotide
- Application of autologous PRFG (Active Comparator): The application of the glues through the external opening of the fistula was controlled by the drainage tube, which was based on fistulography to assure total occlusion of the internal hole. To allow the adhesion of the fibrin glues patch, all fistulous tracts were debrided to produce a smooth surface. At the time of procedures, the two components were mixed together to yield a gelatinous substance. After the FG was instilled, any redundant glue was removed from the external openings.
  Interventions: Procedure: Autologous platelet-rich fibrin glue (PRFG); Drug: Octreotide

INTERVENTIONS:
Procedure: Autologous platelet-rich fibrin glue (PRFG) — 1. Preparation of autologous platelet-rich fibrin glues (PRFG) The platelet-rich plasma (PRP) was separated by centrifugation from 300-400 ml whole blood for 6 min at 1000g, 22°C twice, keeping most of the platelets (50%-60%) in the plasma fraction. For 50g PRP from each patient, with citric acid (2.84mM) lowering and NaHCO3 (75mM) adjusting the PH value, thrombin solution was produced. On the other hand, cryoprecipitate was produced from the rest of the plasma. Frozen at -80°C for at least 6h and then thawed at 4°C, PRP went through centrifugation at 4000rpm/min for 5min.
  2. PRFG application The application of the glues through the external opening of the fistula was controlled by the drainage tube through a double-syringe system with distal mixing device. The distance was based on fistulography to assure total occlusion of the internal hole. After the FG was instilled, any redundant glue was removed from the external openings.
  Arms: Application of autologous PRFG
Drug: Octreotide — subcutaneous injection, 0.3mg/8h until enteral nutrition resolution
  Other Names: Octreotide Acetate Injection, Novartis, Switzerland

SUMMARY:
Adjuvant use of fibrin glue in the fistula tract may promote healing in low-output enterocutaneous fistulas. However, there are only few studies that report autologous glue application in a larger patient group or clinical-controlled studies in this setting. The aim of this study was to investigate the efficacy and safety of autologous platelet-rich fibrin glue (PRFG) in the treatment of low-output digestive fistulas and compare them with conservative management without the use of adjuvant application of FG into the fistulous tract.

DETAILED DESCRIPTION:
The sudden appearance of intestinal contents draining from an abdominal incision is an emotionally devastating experience for both patients and surgeons. An enterocutaneous fistulas (ECF) is an abnormal communication between the bowel lumen and skin, often associated with fluid and electrolyte abnormalities, malnutrition, and sepsis. It is reported that spontaneous fistula closure rates vary from 15% to 71% after conservative treatment with wound care, control of infection, and nutritional support. Sufficient time should be allotted for the ECF to heal with conservative treatment, which also results in long-term discomfort.

Adjuvant use of fibrin glue (FG) in the fistula tract may promote healing in low-output ECF. Containing high concentrations of human fibrinogen and thrombin, FG have been used extensively in many surgical fields as a biological adhesive system for tissue adhesion or hemostasis. Different types of FG are now employed: commercially produced and homemade autologous adhesives. Currently available FDA-approved commercial products such as Tisseel, Artiss (Baxter, Westlake Village, CA, USA), and Evicel (Johnson & Johnson, Somerville, NJ, USA) are widely used in clinical applications. Risks of infection transmission, allergic reactions, and also the high cost, however, still make autologous FG attractive. Additionally, in comparison with other adhesives, autologous compounds have several advantages in terms of biocompatibility and biodegradation.

The aim of this study was to investigate the efficacy and safety of autologous platelet-rich fibrin glue (PRFG) in the treatment of low-output digestive fistulas and compare them with conservative management without the use of adjuvant application of FG into the fistulous tract.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* presence of one or more fistulas
* fistulas of low-output volume (< 200ml/24h)

Exclusion Criteria:

* failure to meet inclusion criteria
* mental handicap
* extreme thinness
* fistulous tract length < 2 cm
* fistulous tract diameter > 1 cm
* entero-atmospheric fistulas
* Crohn's disease-related fistulas
* any conditions that might impede spontaneous closure of the fistula, such as complex tracts, associated abscesses, residual disease, foreign bodies or distal obstruction
* any conditions that might increase the risk of auto-transfusion, including hypertension, or diabetes; and acquired immune deficiency syndrome (AIDS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
counting time from enrollment or glue application to fistula closure or healing (d) | 1-90 days
  The primary measures were defined as the time required for fistula closure and also fistula healing after the last treatment received if in study group, or since enrollment if in control group. Closure was predefined as the absence of drainage through the external openings whether occurring spontaneously or under externally applied pressure. Healing was predefined as complete reepithelialization of external openings.

SECONDARY OUTCOMES:
counting time from enrollment or glue application to enteral intake (d) | 1-90 days
  For secondary analyses, the time required to resume enteral intake from parenteral nutrition was collected. The hospitalization after enrollment, and also the proportion of patients with recurrence of a healed fistula during 12 months follow-up were evaluated. The incidence of adverse events and severe adverse events (defined as an event that was fatal or life-threatening, led to hospitalization or disability, or required an intervention to prevent one of these outcomes) was determined at each study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wu X, Ren J, Gu G, Wang G, Han G, Zhou B, Ren H, Yao M, Driver VR, Li J. Autologous platelet rich fibrin glue for sealing of low-output enterocutaneous fistulas: an observational cohort study. Surgery. 2014 Mar;155(3):434-41. doi: 10.1016/j.surg.2013.09.001. Epub 2013 Oct 29. PMID 24183344